CLINICAL TRIAL: NCT07155915
Title: Effects of Cherry Consumption on Metabolic Health: A Pilot Clinical Study on Healthy Adults
Brief Title: Effects of Cherry Consumption on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico da Guarda (Other)
Responsible Party: Principal Investigator, Luis Manuel Lopes Rodrigues da Silva, Principal Investigator, Instituto Politécnico da Guarda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRR-C05-i03-I-000143
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Health
Keywords: cherry consumption; metabolic health; phenolic compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily Sweet Cherry Consumption (Experimental): Participants in this arm will consume 280 grams of fresh sweet cherries (Prunus avium, "Prime-Giant" variety) every day for 42 consecutive days.
  Interventions: Dietary Supplement: Sweet cherries, 280 g daily for 42 days

INTERVENTIONS:
Dietary Supplement: Sweet cherries, 280 g daily for 42 days — Participants will consume 280 grams of fresh sweet cherries daily for 42 consecutive days. Cherries are provided in pre-weighed portions to be consumed in the morning on an empty stomach

SUMMARY:
This study is designed to evaluate the effects of daily sweet cherry consumption on markers of metabolic health in adults. Cherries are rich in bioactive compounds, such as anthocyanins and phenolic acids, which may help reduce oxidative stress, inflammation, and early risk factors for conditions like type 2 diabetes and cardiovascular disease. Participants will consume 280 grams of fresh sweet cherries every day for 42 consecutive days. Blood and urine samples will be collected at four time points: before the intervention (baseline), at day 21, at day 42 (end of the intervention), and two weeks after stopping cherry consumption.

The study will measure changes in blood sugar regulation, markers of inflammation, oxidative stress, liver and kidney function, and immune response. Waist circumference and body mass index will also be recorded.

The aim of this study is to test whether daily cherry consumption can support metabolic health in healthy adults and to provide data that may inform larger and longer clinical trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Healthy individuals with no known metaboli disorders

Exclusion Criteria:

* Alcohol consumption
* Smoking
* Adverse or allergic reaction to cherries
* Use of antibiotics, anxiolytics, or dietary supplements
* Pregnancy or lactation
* Weight changes greater than 10% in the previous year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Changes in fasting glucose | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in HbA1c | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in estimated average glucose | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in insulin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in IL-6 | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in AGP-1 | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in C-reactive protein | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in gluthatione peroxidase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in gluthatione reductase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in glutamate dehydrogenase | Baseline, Day 21, Day 42 and 2 weeks post-intervention

SECONDARY OUTCOMES:
Changes in aspartate aminotransferase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in alanine transaminase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in gamma-glutamyl transferase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in total bilirubin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in conjugated bilirubin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in unconjugated bilirubin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in lactate dehydrogenase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in total proteins | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in albumin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in urea | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in creatinine | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in microalbumin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in uric acid | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in iron | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in TIBC | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in transferrin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in ferritin | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in amylase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in lipase | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in IgA | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in IgG | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in IgM | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in total IgE | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in rheumatoid factor | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in antistreptolysin O | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in triglycerides | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in total cholesterol | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in HDL cholesterol | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in LDL cholesterol | Baseline, Day 21, Day 42 and 2 weeks post-intervention
Changes in waist circumference | Baseline and Day 42
Body Mass Index | Baseline and Day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Politécnico da Guarda, Guarda, Portugal

IPD SHARING:
Plan to Share IPD: No